CLINICAL TRIAL: NCT00414518
Title: An Open-Label Randomized Clinical Trial to Evaluate the Efficacy and Safety of Short Course Antiretroviral Therapy for Acute or Recent HIV-1 Infection in Zimbabwe and the United States
Brief Title: Safety and Effectiveness of Short-Term Anti-HIV Drug Therapy for Recent HIV-1 Infection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 06-0757; P01AI055356 (NIH); NCT00525070 (obsolete NCT alias); NCT01030172 (obsolete NCT alias)
Record Dates: First submitted 2006-12-19; First posted 2006-12-21 (Estimated); Results first posted 2013-02-20 (Estimated); Last update posted 2013-02-20 (Estimated); Status verified 2013-01

CONDITIONS: HIV Infections
Keywords: Acute Infection; Early HIV Infection; Short-Term Antiretroviral Therapy; Treatment Interruption; Antiretroviral Drug (ARV); ART
MeSH Terms: conditions — HIV Infections | interventions — Tenofovir; Emtricitabine; Lopinavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment interruption (Experimental): Oral Tenofovir disoproxil fumarate/Emtricitabine and Lopinavir/Ritonavir for 12 weeks followed by treatment interruption if CD4 count is 450 mm^3 or higher. When CD4 count is less than 350 mm^3 on two separate, consecutive measurements during treatment interruption, therapy will be resumed.
  Interventions: Drug: Tenofovir disoproxil fumarate/Emtricitabine; Drug: Lopinavir/Ritonavir
- CD4 T cell guided therapy (Experimental): Anti Retroviral Therapy initiated when AIDS-defining illness occurs or if CD4 count is confirmed at less than 350 mm^3 at two separate, consecutive measurements
  Interventions: Drug: Tenofovir disoproxil fumarate/Emtricitabine; Drug: Lopinavir/Ritonavir

INTERVENTIONS:
Drug: Tenofovir disoproxil fumarate/Emtricitabine — 300 mg Tenofovir disoproxil fumarate/ 200 mg emtricitabine tablet taken orally once daily
  Other Names: TDF/FTC
Drug: Lopinavir/Ritonavir — Three 400 mg lopinavir/ 100 mg ritonavir soft gel capsules taken orally twice daily
  Other Names: LPV/RTV

SUMMARY:
The purpose of this study is to determine the safety and effectiveness of an anti-HIV drug regimen followed by treatment interruption in people recently infected with HIV. This study will also compare the effects of a treatment regimen including treatment interruption with a treatment plan based on clinical indicators.

DETAILED DESCRIPTION:
About 6 months after infection, HIV viral load reaches a temporarily stable level known as virus set point. Virus set point is different for each patient and can be a predictor for disease progression. Preliminary studies indicate that early, short-term antiretroviral therapy (ART) given to people newly infected with HIV may lead to lower virus set points and preserved CD4 counts. However, the length of short-term treatment needed to balance the possible adverse effects of ART with the achievement of lower virus set point is not yet known. By lowering the virus set point and maintaining CD4 counts, the need for long-term ART may be postponed. The purpose of this study is to determine the safety and efficacy of a short course of ART on producing a lower virus set point in adults recently infected with HIV.

This study will last at least 28 weeks. Participants will be randomly assigned to one of two arms. Arm A will receive ART for 12 weeks as emtricitabine/tenofovir disoproxil fumarate (TDF/FTC) daily and lopinavir/ritonavir (LPV/RTV) in tablet form twice daily. After 12 weeks, treatment will be interrupted unless the CD4 count is measured to be less than 350 cells/mm^3 on two consecutive occasions during treatment interruption. If that occurs therapy will be resumed. Participants in Arm B will receive no treatment until cluster of differentiation 4 (CD4) counts drop below 350 cells/mm^3, indicating ART is needed. Study visits will occur at study entry, at Weeks 2 and 4, and every 4 weeks thereafter. At each study visit, a physical exam, blood collection, and completion of an adherence questionnaire will occur. Participants are encouraged to enroll in a related substudy that will evaluate HIV viral load in genital secretions.

ELIGIBILITY:
Inclusion Criteria:

* Acute or recent HIV-1 infection. More information about this criterion can be found in the protocol.
* CD4 count 500 cells/mm3 or greater
* No evidence of prior or current AIDS-defining illness
* No signs or symptoms of HIV infection or AIDS-defining illness that, in the opinion of the investigator, requires ART
* Willing to use acceptable forms of contraception

Exclusion Criteria:

* Prior treatment with any antiretroviral drug for more than 7 days
* Use of certain drugs within 21 days of study entry
* Prior receipt of investigational anti-HIV-1 vaccine
* Ongoing therapy with systemic corticosteroids, chemotherapeutic agents, nephrotoxic systemic agents, immunomodulatory treatments, or investigational agents
* Known allergy/sensitivity to study drugs or their formulations
* Current drug or alcohol use or abuse that, in the opinion of the investigator, may interfere with the study
* Serious medical or psychiatric illness that may interfere with the study
* Hepatitis B infected
* Pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2007-01; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michelle A. Barron, MD, Study Chair — Division of Infectious Disease, University of Colorado Health Sciences Center; Margaret Borok, MRCP, Study Chair — Department of Medicine, University of Zimbabwe
Locations (3):
- United States (2):
  - University of Colorado Health Sciences Center, Denver, Colorado
  - AIDS Research Consortium of Atlanta, Atlanta, Georgia
- University of Zimbabwe College of Health Sciences, Harare, Zimbabwe

REFERENCES:
- [Background] Altfeld M, Rosenberg ES, Shankarappa R, Mukherjee JS, Hecht FM, Eldridge RL, Addo MM, Poon SH, Phillips MN, Robbins GK, Sax PE, Boswell S, Kahn JO, Brander C, Goulder PJ, Levy JA, Mullins JI, Walker BD. Cellular immune responses and viral diversity in individuals treated during acute and early HIV-1 infection. J Exp Med. 2001 Jan 15;193(2):169-80. doi: 10.1084/jem.193.2.169. PMID 11148221
- [Background] Fidler S, Oxenius A, Brady M, Clarke J, Cropley I, Babiker A, Zhang HT, Price D, Phillips R, Weber J. Virological and immunological effects of short-course antiretroviral therapy in primary HIV infection. AIDS. 2002 Oct 18;16(15):2049-54. doi: 10.1097/00002030-200210180-00010. PMID 12370504
- [Background] Coombs RW, Speck CE, Hughes JP, Lee W, Sampoleo R, Ross SO, Dragavon J, Peterson G, Hooton TM, Collier AC, Corey L, Koutsky L, Krieger JN. Association between culturable human immunodeficiency virus type 1 (HIV-1) in semen and HIV-1 RNA levels in semen and blood: evidence for compartmentalization of HIV-1 between semen and blood. J Infect Dis. 1998 Feb;177(2):320-30. doi: 10.1086/514213. PMID 9466517
- [Background] Gallant JE. Current status of antiretroviral treatment interruption and intermittent therapy strategies. MedGenMed. 2002 Sep 19;4(3):19. No abstract available. PMID 12466762
- [Background] Gulick RM. Structured treatment interruption in patients infected with HIV: a new approach to therapy. Drugs. 2002;62(2):245-53. doi: 10.2165/00003495-200262020-00001. PMID 11817971

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment Interruption: Oral tenofovir/emcitribine (TDF/FTC) and lopinavir/ritonavir(LPV/RTV) for 12 weeks followed by treatment interruption if CD4 count is 450 mm^3 or higher. When CD4 count is less than 350 mm^3 on two separate, consecutive measurements during treatment interruption, therapy will be resumed.
- CD4 T Cell Guided Therapy: Antiretroviral therapy (ART) will not be initiated until AIDS-defining illness occurs or if CD4 is confirmed at less than 350 mm^3 at two separate, consecutive measurements
Period: Overall Study
Arm/Group | Treatment Interruption | CD4 T Cell Guided Therapy
Started | 7 | 9
Completed | 7 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Arm A: Oral tenofovir/emcitribine (TDF/FTC) and lopinavir/ritonavir(LPV/RTV) for 12 weeks followed by treatment interruption if CD4 count is 450 mm^3 or higher. When CD4 count is less than 350 mm^3 on two separate, consecutive measurements during treatment interruption, therapy will be resumed.
- Arm B: Antiretroviral therapy (ART) will not be initiated until AIDS-defining illness occurs or if CD4 is confirmed at less than 350 mm^3 at two separate, consecutive measurements
- Total: Total of all reporting groups
Arm/Group | Arm A | Arm B | Total
Number analyzed (Participants) | 7 | 9 | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 9 | 16
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 8
  Male | 4 | 4 | 8
Region of Enrollment [Number; unit: participants]
  United States | 3 | 4 | 7
  Zimbabwe | 4 | 5 | 9

OUTCOME MEASURES:

1. Primary Outcome: Plasma HIV-1 Viral Load (Copies/ml) at Week 24 as Compared Between the Two Arms
Time Frame: At Week 24
Measure: Mean (Standard Deviation); unit: Log 10 copies of virus/ml
Groups:
- 12 Week Treatment Arm Followed by Treatment Interruption: Oral tenofovir/emcitribine (TDF/FTC) and lopinavir/ritonavir(LPV/RTV) for 12 weeks followed by treatment interruption if CD4 count is 450 mm^3 or higher. When CD4 count is less than 350 mm^3 on two separate, consecutive measurements during treatment interruption, therapy will be resumed.
- CD4 T Cell Guided Therapyh: Antiretroviral therapy (ART) will not be initiated until AIDS-defining illness occurs or if CD4 is confirmed at less than 350 mm^3 at two separate, consecutive measurements
Arm/Group | 12 Week Treatment Arm Followed by Treatment Interruption | CD4 T Cell Guided Therapyh
Number analyzed (Participants) | 7 | 9
Log 10 copies of virus/ml | 4.8627 (0.9055) [infinity to 1.5] | 4.2620 (1.0867) [infinity to 1.37]

2. Primary Outcome: Number of Participants Experiencing Either an AIDS-defining Event, a Grade 3 or 4 Adverse Event, or Acute Retroviral Syndrome
Time Frame: At Week 24
Measure: Number; unit: participants
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 7 | 9
participants | 1 | 1

3. Primary Outcome: Viral Set Point
Description: set point is reached after the immune system has developed HIV antibodies and begins to attempt to fight the virus
Time Frame: Throughout study
Measure: Mean (Standard Deviation); unit: Log 10 copies virus/ml
Groups:
- 12 Week Treatment Folllowed by Treatment Interruption: Oral tenofovir/emcitribine (TDF/FTC) and lopinavir/ritonavir(LPV/RTV) for 12 weeks followed by treatment interruption if CD4 count is 450 mm^3 or higher. When CD4 count is less than 350 mm^3 on two separate, consecutive measurements during treatment interruption, therapy will be resumed.
Arm/Group | 12 Week Treatment Folllowed by Treatment Interruption | CD4 T Cell Guided Therapy
Number analyzed (Participants) | 7 | 9
Log 10 copies virus/ml | 4.8627 (0.9055) | 4.2434 (0.7992)

ADVERSE EVENTS:
Arm/Group | Arm A | Arm B
Serious Adverse Events (participants affected / at risk) | 1/7 | 1/9
Other Adverse Events (participants affected / at risk) | 3/7 | 5/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (N=7) | Arm B (N=9)
grade 3 abnormal serum phosphorous level (Metabolism and nutrition disorders) | 1 (2) | 0 (0) — One patient randomized to Arm A experienced a grade 3 abnormal serum phosphorous level at week 4 and 16. The adverse event was not treatment limiting.
grade 3 headache (Nervous system disorders) | 0 (0) | 1 (1) — One subject randomized to Arm B experienced a grade 3 headache at baseline. The adverse event was not treatment limiting.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (N=7) | Arm B (N=9)
low absolute neutrophil count (ANC) (Blood and lymphatic system disorders) | 3 (3) | 4 (4)
Elevated aspartate amino transferase (Metabolism and nutrition disorders) | 1 (1) | 5 (5)
abnormal hemoglobin (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
abnormal phosphorus (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
ache/pain/discomfort (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (4)
abnormal alanine amino transferase (Metabolism and nutrition disorders) | 1 (1) | 3 (3)
abnormal glucose (Endocrine disorders) | 3 (3) | 0 (0)
fatigue/malaise (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
fever (Infections and infestations) | 2 (2) | 1 (1)
headache (Nervous system disorders) | 1 (1) | 1 (1)
abnormal uric acid (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
congestion/effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
abnormal sodium (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
blister/ulcer/lesions (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
chills/rigors/sweats/night sweats (Infections and infestations) | 0 (0) | 1 (1)
constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
abnormal fasting blood sugar (Endocrine disorders) | 1 (1) | 0 (0)
macules/papules/rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
mucous membrane/skin abnormality (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
nausea and vomiting/vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
weakness (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No